CLINICAL TRIAL: NCT01667601
Title: The Effectiveness of a Mindfulness-based Illness Management Program for Chinese Patients With Schizophrenia: An Randomised Controlled Trial
Brief Title: Mindfulness-based Illness Management Program for Schizophrenia
Acronym: MBPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government); Jilin Medical College, China (Unknown); Taipei Medical University, Taiwan (Unknown)
Responsible Party: Principal Investigator, Wai-Tong Chien, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20121211001
Record Dates: First submitted 2012-08-15; First posted 2012-08-17 (Estimated); Last update posted 2019-12-18 (Actual); Status verified 2017-07

CONDITIONS: Schizophrenia
Keywords: mindfulness-based program; Psychoeducation; schizophrenia; Chinese; outpatients
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Mindfulness-based program (Experimental): A structured, researcher-designed mindfulness-based psycho-education program (6 months), comprised of 12 bi-weekly, 2-hour group sessions (10-12 patients per group). The program was based on the psycho-education programs by Chien et al. (2010) and Lehman et al. (2004), as well as the 8-session Mindfulness-Based Stress Reduction Program by Kabat-Zinn (1990).
  Interventions: Behavioral: Mindfulness-based program
- Routine Care (Other): Routine psychiatric outpatient care, including medication, psychiatric consultation in outpatient clinic, brief education by psychiatric nurses, financial and social welfare advices by social workers, and individual counseling by clinical psychologist.
  Interventions: Other: Routine Care; Behavioral: Mindfulness-based program; Behavioral: Psychoeducation group
- Psychoeducation group (Active Comparator): A psychoeducation group program (12 sessions, bi-weekly) based on Dr. Macpherson's Family Psychoeducation Program in 1996 and Chien and Bressington's one in 2014/15 will be used.
  References:
  Chien WT, Bressington D. A randomized controlled trial of a nurse-led structured psychosocial intervention program for people with first-onset mental illness in psychiatric outpatient clinics. Psychiatry Res 2015;229:277-86.
  Macpherson R, Jerrom B, Hughes AA. controlled study of education about drug treatment in schizophrenia. Br J Psychiatry 1996;168:709-17.
  Interventions: Behavioral: Psychoeducation group

INTERVENTIONS:
Other: Routine Care — Psychiatric outpatient care provided by the outpatient departments, e.g., medical consultation, brief education by psychiatric nurses and financial advices or referrals by social workers.
  Other Names: Routine Psychiatric Care
  Arms: Routine Care
Behavioral: Mindfulness-based program — The program was based on the psychoeducation programs by Chien et al and Lehman et al, as well as the 8-session Mindfulness-Based Stress Reduction Program by Kabat-Zinn(1990).
  Other Names: Mindfulness-based illness management program; Mindfulness-based care for schizophrenia program
  Arms: Mindfulness-based program; Routine Care
Behavioral: Psychoeducation group — A 5-month patient psychoeducation group program (12 sessions) led by the research team will be provided.
  Other Names: Conventional psychoeducation group; Psychoeducation group intervention
  Arms: Psychoeducation group; Routine Care

SUMMARY:
Only a few intervention studies have also focused on changing patients' negative thoughts and feelings towards the illness and their relationship to the suffering caused by those thoughts, which is evidenced to empower psychosocial functioning and control of distressing thoughts in severe depression and psychotic disorders by using the Mindfulness-Based Stress Reduction program. This controlled trial is designed to test the effects of a mindfulness-based Illness management program (MBPP) for Chinese patients with schizophrenia on their symptom severity, illness insight and psychosocial functioning.

DETAILED DESCRIPTION:
Objectives: This study is to test the effectiveness of a mindfulness-based illness management program for Chinese outpatients with schizophrenia over a 24-month follow-up. The program is an integrated, insight-inducing educational program that addresses patients' awareness and knowledge of schizophrenia and skills of illness management.

Methods: A two-phase, single-blind, multi-site randomized controlled trial will be conducted with 449 Chinese patients with schizophrenia in Hong Kong, China and Taiwan. In the first phase, 107 participants will be randomly selected from the eligible patient lists of three outpatient clinics in Hong Kong only (i.e., 38 subjects from each clinic), and after baseline measurement, be assigned to either the mindfulness-based illness management program, conventional psycho-education group, or usual psychiatric care. For the second phase, the participants will be randomly selected from the eligible patient list in three study venues or countries (i.e., 114 subjects from each study site/ country) and after baseline measurement, be assigned similar to the first phase to one of the three study groups. The patients' mental and psychosocial functioning, insights into illness, and their re-hospitalization rates will be measured at recruitment and at one week, and 6, 12 and 24 months after completing the interventions.

Hypothesis: The patients in the mindfulness-based psycho-education program will report significantly greater improvements in their symptoms and re-hospitalization rates (primary outcomes) and other secondary outcomes (e.g., insight into illness and functioning) over the 24-month follow-up, when compared with those in psycho-education group or usual care.

Conclusions: The findings will provide evidence whether the mindfulness-based psycho-education program can better improve Chinese schizophrenia sufferers' psychosocial functioning and reduce their illness relapse.

ELIGIBILITY:
Inclusion Criteria:

* outpatients;
* aged 18+; and
* diagnosed as schizophrenia and other psychotic disorders (< or =5 years) according to the Diagnostic and Statistical Manual, 4th edition, as ascertained by the Structured Clinical Interview (SCID-I).

Exclusion Criteria:

* not able to understand the psycho-education content and Chinese;
* mentally unstable at recruitment; and
* with co-morbidity of other severe mental health problems such as depression and substance misuse.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 449 (Actual)
Dates: Start 2010-08; Primary Completion 2016-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Rehospitalization rates | from recruitment to 24-month follow-up
  Average amount (number) and length of hospital stay of the patients over previous six months will be assessed at recruitment and one week, 6 months, 12 months and 24 months after the interventions completed.
Positive and Negative Syndrome Scale | from recruitment to 24-month follow-up
  The Positive and Negative Syndrome Scale assesses the severity of psychotic symptoms on three subscales: positive symptoms (7 items), negative symptoms (7 items) and general psychopathology (16 items). will be assessed at recruitment and one week, 6 months, 12 months and 24 months after the interventions completed. Symptom remission rate over the follow-up periods are also assessed. Complete remission was defined as 4-month simultaneous ratings of all individual items in PANSS as score ≤3.

SECONDARY OUTCOMES:
insights to illness and treatment | from recruitment to 24-month follow-up
  Patients' insight and attitudes to illness and treatment will be measured with the Insight and Treatment Attitudes Questionnaire at recruitment and one week, 6 months, 12 months and 24 months after the interventions completed.

OTHER OUTCOMES:
Specific Level of Functioning Scale | from recruitment to 24-month follow-up
  Patients' levels of psychosocial functioning will be assessed with the Specific Level of Functioning Scale at baseline and one week, 6 months, 12 months and 24 months follow-up.
Six-item Social Support Questionnaire | from recruitment to 24-month follow-up
  Patients' perceived social support will be assessed with the Six-item Social Support Questionnaire at baseline and one week, 6 months, 12 months and 24 months follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Chien WT, PhD, Principal Investigator — The HK Polytechnic University
Locations (4):
- Jilin Medical College, Jilin, Jilin, China
- Hong Kong (2):
  - KH/LKS Specialty OPD, Shatin, NT
  - TM Psy Centre, Tuenmen, NT
- Taipei Medical University, Taipei, Xinyi, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chien WT, Lee IY. The mindfulness-based psychoeducation program for Chinese patients with schizophrenia. Psychiatr Serv. 2013 Apr 1;64(4):376-9. doi: 10.1176/appi.ps.002092012. PMID 23412024
- [Background] Chien WT, Thompson DR. Effects of a mindfulness-based psychoeducation programme for Chinese patients with schizophrenia: 2-year follow-up. Br J Psychiatry. 2014 Jul;205(1):52-9. doi: 10.1192/bjp.bp.113.134635. Epub 2014 May 8. PMID 24809397
- [Background] Lam, A.H.Y., & Chien, W.T. (2016). The effectiveness of mindfulness-based intervention for people with schizophrenia: A systematic review. Neuropsychiatry (London), 6(5), 208-222.
- [Result] Chien WT, Bressington D, Yip A, Karatzias T. An international multi-site, randomized controlled trial of a mindfulness-based psychoeducation group programme for people with schizophrenia. Psychol Med. 2017 Sep;47(12):2081-2096. doi: 10.1017/S0033291717000526. Epub 2017 Apr 4. PMID 28374661